CLINICAL TRIAL: NCT01547234
Title: Observational Study for Assessment of the Effect of Fampyra on the Manual Function of Persons With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ariel Miller, Director of Multiple Sclerosis & Brain Research Center, Carmel Medical Center
Other Study IDs: CMC-11-0081-CTIL; FAM-MS-2011 (Registry Identifier: Fampyra)
Record Dates: First submitted 2012-02-23; First posted 2012-03-07 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; ambulation; manual function; Fampridine
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Multiple Sclerosis (MS) is the most common chronic neurological disease affecting young adults, with onset usually at age 20-40 years. Women are affected 3-4 times more than men. The disease is characterized by 2 main phenotypes: relapsing-remitting or progressive course.

Several immunotherapies were developed in the last 10-15 years for the long term management of the relapsing type of disease. Treatment with these drugs decreases disease activity though cannot cure it.

There are few treatments for targeting specific symptoms of MS, such as Provigil for the treatment of fatigue.

Regarding problems related to spasticity and related gait problems , which is stated by over 40 % of MS patients as their main complaint - present treatments include: non-pharmacological treatments such as physiotherapy, occupational therapy, hydrotherapy and pharmacological treatments such as Baclofen, Tizanidine and Botulinium toxin.

Fampyra (Fampridine) has recently been approved for use in patients with gait problems. This drug acts by blocking potassium ion channels and has been proven to improve walking in 35% of the patients after one month of treatment.

The effect of Fampyra on hand function in MS has yet to be studied. The aim of this research project is to assess the effect of treatment with Fampyra on manual function of patients with MS. The investigators hypothesize that through the same mechanism by which Fampyra improves ambulation it can also improve manual function.

MS patients visiting the MS center clinic at the Carmel Medical Center, with walking disabilities eligible to Fampyra treatment, that have also manual dysfunction, will be offered to participate in this study. Participants who agree to participate will be asked to sign a written informed consent. Information regarding their personal and family medical history will be collected via questionnaires. Medical staff will fill clinical questionnaires detailing patient clinical status prior to the study.

Patients will be followed up to 4 months after initiation of treatment with Fampyra. Compliance to treatment will be assessed by collection of the empty vials of the medication.

In each of the follow-up meetings evaluation of manual function, evaluation of ambulation and evaluation of general neurological function will be performed.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE Multiple Sclerosis (MS) is the most common chronic neurological disease affecting young adults, with onset usually at age 20-40 years. Women are affected 3-4 times more than men. The disease is characterized by 2 main phenotypes: relapsing-remitting or progressive course.

Relapsing-remitting (RR) MS is the most common type of disease, affecting 60 to 85% of the patients. This form is characterized by relapses that lead to disability followed by periods of remission that may last for month to decades. During remission patients experience a significant improvement in their condition.

This form may transform into another disease type: Secondary progressive (SP) MS, in which there is a continuous deterioration in disability between relapses.

Primary-progressive (PP) MS- is characterized by a progressive decline in the patient condition with no remission.

MS is a complex multi-factorial disease, with underlying both genetic and environmental factors. Different populations have different susceptibility. It is characterized by the invasion of cells of the immune system cells into the central nervous system (CNS) provoking an inflammatory reaction against the myelin -producing cells- the olgodendrocytes as well as neurodegeneration. Myelin is an electrically insulating material that surrounds the axon and enhances the passage of electrical signals within the CNS.

As a consequence of these neuro-inflammatory and neurodegenerative processes in the CNS, a the various neurologic systems may be affected: motor, sensory, visual, cognitive cerrebellar and sphincters,, leading to a variety of neurological symptoms and signs, accordingly.

Treatment: Following the increased understanding of the disease in the last 10-15 years, subcutaneous injection immunotherapies available for the long term management including Glatiramer acetate- copaxon and interferon beta derivatives- Avonex, Rebif, and Betaferon , and Tysabri were developed and approved for treatment. An orally administered drug has been recently approved for use - Gilenya, and others are currently being developed.

Treatment with these drugs decreases disease activity, though cannot cure the disease. These treatments are only partially efficient and are suitable only for patients with RRMS. There is no available treatment for patients with PPMS whose disability progresses continuously over time.

In addition to disease modifying therapies (DMTs) which are immunomodulatory for controlling disease activity and progression, there are few treatments for targeting specific symptoms of MS, such as: Provigil for the treatment of fatigue.

Regarding problems related to spasticity and related gait problems , which is stated by over 40 % of MS patients as their main complaint - present treatments include: non-pharmacological treatments such as physiotherapy, occupational therapy, hydrotherapy and pharmacological treatments such as Baclofen, Tizanidine and Botulinium toxin.

Fampyra (Fampridine) has recently been approved for use in patients with gait problems. This drug acts by blocking potassium ion channels and has been proven to improve walking in 35% of the patients. Improvement can be seen after one month of treatment. Presently, this medication is offered to all MS patients with walking disabilities as it cannot be predicted which patients will benefit from it.

The most common adverse reactions are: Urinary tract infection, Insomnia, Dizziness, Headache, Nausea, Asthenia, Back pain.

Less common adverse reaction: MS relapse, Paresthesia, Nasopharyngitis, Constipation, Dyspepsia, Pharyngolaryngeal pain.

In addition, in high doses (> 10mg two times a day) the drug increases the risk for seizures and is therefore contraindicated in patients with moderate-severe renal failure and history of seizure.

Fampyra was approved for the treatment of walking disabilities in MS patients but the effect of Fampyra on hand functions in MS has yet to be studied. Since Fampyra improves walking functions in persons with MS by blocking potassium channels and therefore improving nerve conductivity, it may also affect hands functions through the same mechanism.

The aim of this research project is to assess the effect of treatment with Fampyra on hands functions of patients with MS.

PATIENTS RECRUITMENT MS patients visiting the MS center clinic at the Carmel Medical Center, with walking disabilities eligible to Fampyra treatment, that have also manual dysfunction, will be offered to participate in this study. Participants will receive an explanation from Prof. Miller, or the attending neurologist authorized by Prof Miller to do so, on the study aims and protocol, and sign an informed consent. Information regarding their personal and family medical history, including data such as education and occupation, demographic and ethnicity data, data on smoking and diet habits will be collected via questionnaires. Medical staff will fill clinical questionnaires detailing patient clinical status prior to the study. Data will also be collected from medical records, as necessary. Data collected through participants and physician filled forms and from medical records will be stored in an Excel data base. The medication will be provided in line with the indication in the Israeli health basket.

FOLLOW UP PROGRAM Meetings' schedule

1. 2-4 weeks before starting the Fampyra treatment.
2. A month after starting the Fampyra treatment.
3. 3 months after starting the Fampyra treatment.
4. 4 months after starting the Fampyra treatment.

Compliance to treatment will be assessed by collection of the empty vials of the medication.

In each of the 4 meetings the following evaluations will be performed:

I. Evaluation of manual function:

1. Computerized Penmanship Evaluation Tool (ComPET) - An objective evaluation tool, including digitizing tablet and on-line handwriting data collection and analysis software.This unique data collection and analysis program including a suite of on-line, computerized tasks programmed in C++ and implemented via MATLAB software toolkits, was used to administer the stimuli and to collect and analyze the data. The writing tasks were performed on A4 size lined paper (spacing=0.5 cm) affixed to the surface of a WACOM Intuos II (407 X 417 X 36.3 mm) x-y digitizing tablet using a wireless electronic pen with a pressure sensitive, inking tip (model Up 401). The pen size and weight are similar to those of a normal pen (length=150 mm, circumference=35 mm, weight=11 gm). Displacement, pressure, and pen tip angle were sampled at 100 Hz via a 90 MHz Pentium laptop computer. Writing tasks include the participant's signature and the copying of a short paragraph. The rational for the selection of these items was that both of them are commonly occurring functional tasks that have relevance for the participant. Signing one's signature is more familiar and is hence executed almost automatically. Copying a short paragraph is somewhat more complex and lengthy and would thus reflect every day performance during prolonged tasks that entail perceptual-motor components and integration.

   The system samples temporal, spatial and pressure data. The outcome measures, based on previous study results and the known characteristics of patients with MS, included On-paper and In-air time (i.e., the time while writing in which the pen is not in contact with the paper in seconds) for the whole task or for each segment, mean segment width and length in millimeters, and mean pressure and mean standard deviation of pressure in non-scaled units from 0-1023. This computerized system enables dynamic handwriting evaluation; previous studies established the ComPET's discriminate validity between control group and groups of participants with varied pathologies as well as between age groups. Concurrent validity was also established.

   The writing text will be in the Hebrew, Russian and Arabic language according to patient preference.

   The text that the participants would be requested to copy annexed in appendix 1.
2. Nine Hole Peg test - This is a simple test to evaluate coordination and fine motor skills which has been proven reliable in previous studies. This is a timed test where the patient must insert nine small pegs into nine corresponding holes.
3. Arthritis Hand Function test - This test comprehends a list of daily activities tests. Patients will perform 5 tasks: shoelace tying, fastening/unfastening 2 safety pins, pouring a glass of water, buttoning and inserting coins into a container. Activities will be timed and a score will be given accordingly.
4. Jamar Dynamometer - This apparatus serves to document manual function by measuring the grip strength. It is based on hydraulics and measures isometric strength. It has been proven in previous studies to be reliable and safe.
5. Pinch Meter - In this test the apparatus is held between two fingers (thumb and index) and measures the pinch strength in the hand. It is an useful tool for the early detection of motor function loss.
6. Dreiser Functional Index - This is a ten-question questionnaire which evaluates aspects of daily manual function such as holding cutlery, buttoning, opening locks with keys, etc. This questionnaire is widely used to evaluate the manual function of patients with osteoarthritis.

II. Evaluation of ambulation:

Since Fampyra has been shown to improve walking in about 35% of patients, in participants with both walking disabilities and hand function disabilities, improvement in hand function will be compared to improvement in walking.

As stated earlier, this medication is effective for treatment of mobility problems in only 35% of the patients. Therefore the investigators will evaluate walking improvement and compare it to improvement in hand function.

1. Timed 25-foot walk - This test assesses walking speed. It was used to measure improvement in ambulation in the clinical trials of Fampyra.
2. 12MSWS questionnaire - a 12-question questionnaire specifically designed to assess ambulation in MS patients.

III. General function and questionnaires:

1. General neurological function including Expanded Disability Status Scale (EDSS).
2. Mini-Mental State Exam.
3. Geriatric Depression Scale.
4. Daily Living Questionnaire.
5. Personal, familial and writing characteristics questionnaire.
6. Diagnostic and clinical history questionnaire.
7. Follow up and clinical history questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females diagnosed with Multiple Sclerosis.
2. Over age 18.
3. Walking disabilities and manual dysfunction.
4. Willing and able to give inform consent

Exclusion Criteria:

1. Additional CNS co-morbidity.
2. Renal failure.
3. MS relapse within previous 60 days.
4. History of epilepsy or epileptic brain activity on EEG or other conditions which could affect the interpretation of results.
5. Clinical problems that cause manual disability in addition to MS.

WITHDRAWAL CRITERIA

1. Participants who decide to withdraw from the study for any reason.
2. Pregnancy.
3. Technical problems in performing the tests.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MS patients visiting the Multiple Sclerosis Clinic at the Carmel Medical Center, Haifa
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Score of hand function tests | 1,3,4 months after treatment initiation
  Scores of hand function tests before treatment with Fampyra and at several timepoints after treatment initiation will be compared.

SECONDARY OUTCOMES:
Improvement in daily function | 1,3,4 months after treatment initiation
  Assessment of daily function before treatment with Fampyra and 4 months after initiation of treatment will be compared.
Correlation between improvement in manual function and ambulation | 1,3,4 months after treatment initiation
  Improvement in patient manual function after 1 to 4 months of initiation of treatment with Fampyra will be compared to patient improvement in ambulation over the same period of time.

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Miller, MD,Ph.D, Principal Investigator — Multiple Sclerosis Center Carmel Medical Center
Locations (1):
- Multiple Sclerosis Center Carmel Medical Center, Haifa, Israel